CLINICAL TRIAL: NCT03957720
Title: The Individual Therapy for Patients With Wilson's Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: WuZYLab-WD
Record Dates: First submitted 2019-04-08; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Unithiol; Penicillamine; Succimer; gluconic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- homo-R778L (Experimental): When patients carrying homo-R778L mutation are in hospital, they receive DMPS treatment. Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days; When being off hospital, they receive DMSA treatment. Adult patient,Dosage Form: DMSA: 750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Pediatric patient,Dosage Form: DMSA: 35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Interventions: Drug: DMPS; Drug: DMSA
- R778L+truncation mutation (Experimental): When patients carrying R778L and truncation mutation are in hospital, they receive DMPS treatment.
  Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days; When being off hospital, they receive DMSA treatment. Adult patient,Dosage Form: DMSA: 750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Pediatric patient ,Dosage Form: DMSA: 35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Interventions: Drug: DMPS; Drug: DMSA
- Homo-P992L (Experimental): When patients carrying Homo-P992L mutation are in hospital, they receive DMPS treatment.
  Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days; When being off hospital, they receive DMSA treatment. Adult patient,Dosage Form: DMSA: 750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Pediatric patient ,Dosage Form: DMSA: 35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Interventions: Drug: DMPS; Drug: DMSA
- P992L+truncation mutation (Experimental): When patients carrying P992L and truncation mutation are in hospital, they receive DMPS treatment.
  Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days; When being off hospital, they receive DMSA treatment. Adult patient,Dosage Form:DMSA:750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Pediatric patient,Dosage Form:DMSA:35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Interventions: Drug: DMPS; Drug: DMSA
- T935M+other point mutations (Experimental): When patients carrying T935M and other point mutations are in hospital, they randomly receive DMPS or penicillamine treatment; Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days; Dosage Form: penicillamine: 250-1500mg per day, Frequency:TID,Duration: 5 years; When being off hospital, they receive DMSA treatment or penicillamine. Adult patient,Dosage Form: DMSA: 750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Pediatric patient,Dosage Form: DMSA: 35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Interventions: Drug: DMPS; Drug: Penicillamine; Drug: DMSA
- Presymptomatic patients with Wilson's disease (Experimental): According to different age group, they receive various dosage of Zinc Gluconate treatment.
  Patient aged≤6 years,Dosage Form: Zinc Gluconate: 140mg once, Zinc Gluconate Frequency:BID, Zinc Gluconate Duration: 5 years; Patient aged from 6 to 14 years,Dosage Form: Zinc Gluconate: 140mg once, Zinc Gluconate Frequency:TID, Zinc Gluconate Duration: 5 years; Patient aged≥14 years,Dosage Form: Zinc Gluconate: 210mg once, Zinc Gluconate Frequency:TID, Zinc Gluconate Duration: 5 years;
  Interventions: Drug: Zinc gluconate

INTERVENTIONS:
Drug: DMPS — Dosage Form: DMPS: 500-1000mg per day,DMPS Frequency:BID,DMPS Duration: 6 days;
  Other Names: Sodium Dimercaptosulphonate
  Arms: Homo-P992L; P992L+truncation mutation; R778L+truncation mutation; T935M+other point mutations; homo-R778L
Drug: Penicillamine — Dosage Form: Penicillamine: 250-1500mg per day, Frequency:TID,Duration: 5 years;
  Arms: T935M+other point mutations
Drug: DMSA — Dosage Form: DMSA: 750-1000mg per day,DMSA Frequency:BID,DMSA Duration: 5 years; Dosage Form: DMSA: 35mg/kg per day,DMSA Frequency:BID,DMSA Duration: 5 years;
  Other Names: Dimercaptosuccinic Acid
  Arms: Homo-P992L; P992L+truncation mutation; R778L+truncation mutation; T935M+other point mutations; homo-R778L
Drug: Zinc gluconate — Dosage Form: Zinc gluconate: 140mg per time,Zinc Frequency:BID,Zinc Duration: 5 years; Dosage Form: Zinc gluconate: 140mg per time,Zinc Frequency:TID,Zinc Duration: 5 years; Dosage Form: Zinc gluconate: 210mg per time,Zinc Frequency:TID,Zinc Duration: 5 years;
  Arms: Presymptomatic patients with Wilson's disease

SUMMARY:
Based on the genotype characteristics and genotype-phenotype-treatment prognosis data of Chinese WD patients, this study intends to further optimize the treatment regimen of Chinese WD patients and formulate individualized treatment regimens for each genotype, so as to further improve the prognosis of patients.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate treatment regimen efficacy based on different mutations, and Zinc treatment in presymptomatic WD patients.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Wilson's disease
* Presymptomatic patients with Wilson's disease

Exclusion Criteria:

* Movement disorder due to other definite causes instead of Wilson's disease
* Severe Lung, kidney or liver disease
* Neoplastic Disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum ceruloplasmin | Five years
  Serum ceruloplasmin concentration will be analysed using a validated assay
24-hour urine copper | Five years
  24-hour urinary copper excretion is to be measured
serum copper | Five years
  serum copper will be analysed using a validated assay
White blood cell | Five years
  The white blood cell will be evaluated using a validated assay
Platelet count | Five years
  The platelet count will be evaluated using a validated assay
urine protein level | Five years
  The urine protein level will be collected using a validated assay
Alanine transaminase | Five years
  The concentration of alanine transaminase will be collected using a validated assay
blood creatinine | Five years
  The concentration of blood creatinine will be tested using a validated assay
international normalized ratio | Five years
  The international normalized ratio will be analyzed
hepatic fibrosis markers test | Five years
  The concentrations of procollagen III, collage IV and hyaluronidase will be evaluated using a validated assay
bone mineral density test | Five years
  The bone mineral density will be tested using the dual energy X ray absorptiometry
Abdominal ultrasound | Five years
  The abdominal ultrasound will be collected
Urinary ultrasound | Five years
  The urinary ultrasound will be analyzed in patients
Cranial MRI scan | Five years
  The cranial MRI scan will be analyzed in patients
Unified Wilson's disease rating scale | Five years
  The Unified Wilson's disease rating scale consist of three subscales, including neurological part (0~112), liver functional part (0~36) and mental state part (0~76). Three subscale scores are summed to compute a total score. The higher values represent a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ying Wu, MD&PhD, Principal Investigator — Zhejiang University
Locations (1):
- econd Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No